CLINICAL TRIAL: NCT06830941
Title: Efficacy and Safety of Iron Isomaltoside in the Treatment of Peritoneal Dialysis Patients with Renal Related Anemia: a Randomized Controlled Trial
Brief Title: Iron Isomaltoside for the Treatment of Anemia in Peritoneal Dialysis Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xie Jingyuan, MD (Other)
Collaborators: RenJi Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Songjiang Hospital, Shanghai Jiao Tong University School of Medicine (Unknown); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Chinese People's Liberation Army No 455 Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Xie Jingyuan, MD, professor, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Iron isomaltoside-PD
Record Dates: First submitted 2025-02-10; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Renal Anemia; Peritoneal Dialysis (PD)
Keywords: peritoneal dialysis; renal anemia; iron isomaltoside; iron treatment
MeSH Terms: interventions — iron isomaltoside 1000; ferrous succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Iron isomaltoside Group (Experimental): Intravenous infusion of 1000mg iron isomaltoside as a single dose for over 15min. Iron isomaltoside 1000mg was diluted in 100ml of 0.9% saline.
  Interventions: Drug: Iron isomaltoside
- Ferrous succinate Group (Active Comparator): Patients received ferrous succinate treatment orally given as 200mg twice a day for 8 weeks(containing iron element 7840mg in total).
  Interventions: Drug: Ferrous succinate

INTERVENTIONS:
Drug: Iron isomaltoside — Intravenous infusion of 1000mg iron isomaltoside as a single dose for over 15min. Iron isomaltoside 1000mg was diluted in 100ml of 0.9% saline.
  Other Names: Intravenous iron isomaltoside
  Arms: Iron isomaltoside Group
Drug: Ferrous succinate — Patients received ferrous succinate treatment orally given as 200mg twice a day for 8 weeks.
  Other Names: Oral ferrous succinate
  Arms: Ferrous succinate Group

SUMMARY:
This is a prospective multicenter randomized controlled clinical study. The goal of this clinical trial is to learn if intravenous iron isomaltoside injection use is equally effective and safe for the treatment of renal anemia in peritoneal dialysis patients compared with oral ferrous succinate tablets.

The main questions to answer are:

* Changes in hemoglobin concentration from baseline to week 8 after the use of single dose intravenous iron isomaltoside injection in peritoneal dialysis patients with renal anemia.
* If intravenous iron isomaltoside injection use is equally effective and safe for the treatment of renal anemia in peritoneal dialysis patients compared with oral ferrous succinate tablets.

Participants will:

* be randomized 1:1 to two groups, either Iron isomaltoside Group (Group A, experimental group) or Ferrous succinate Group (Group B, control group).
* Patients in Iron isomaltoside Group will receive a single dose of intravenous iron isomaltoside injection, the dose of which is set at 1000 mg. Patients in Ferrous succinate Group will receive ferrous succinate treatment orally given as 200mg twice a day for 8 weeks (containing iron element 7840mg in total).
* Patients will be followed up for 8 weeks.

DETAILED DESCRIPTION:
This is a prospective multicenter randomized controlled clinical study. The purpose of this study is to evaluate the efficacy and safety of single dose intravenous iron isomaltoside comparing with daily oral ferrous succinate in the treatment of renal anemia among patients on peritoneal dialysis.

A total of 124 patients will be enrolled. The primary endpoint is hemoglobin change from baseline to week 8, the secondary endpoint is hemoglobin change from baseline to week 4. Other secondary endpoints include the results of iron metabolism, reticulocytes, composite cardiovascular events, laboratory and safety parameters. The expected result is that intravenous iron isomaltoside is equally effective and safe for the treatment of renal anemia in peritoneal dialysis patients compared with oral ferrous succinate tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females who are ≥ 18 years and on PD treatment for ≥90 days, body weight≥50Kg
2. Hemoglobin(Hb）≤110 g/L at screening phase
3. Serum ferritin(SF）≤200 μg/L or transferrin saturation(TSAT）≤20% at screening phase
4. No oral or intravenous iron use within 4 weeks prior to screening.
5. No hypoxia-inducible factor prolyl hydroxylase inhibitor（HIF-PHI）used or other erythropoiesis-stimulating agent（ESA）except for erythropoietin (EPO) used in the past 4 weeks prior to screening
6. Stable doses of erythropoiesis-stimulating agents (ESA) with a change of dose ≤20% during the past 4 weeks.
7. Willing to participate and signed the informed consent form

Exclusion Criteria:

1. Anemia predominantly caused by other diseases rather than renal diseases according to the investigator's judgement. (eg. bleeding, hematological diseases, anemia due to autoimmune diseases)
2. History of disturbances in iron utilisation.(eg. hemochromatosis and hemosiderosis）
3. Anemia due to lack of folate or vitamin B12：folate<6.8nmol/L（3ng/ml）and(or) Vitamin B12<74pmol/L（100pg/ml）at screening phase
4. Histories of serious allergies to iron
5. Obvious liver dysfunction：ALT>3×ULN and/or AST>3×ULN，or total bilirubin>1.5×ULN
6. Active acute or chronic infection(clinically diagnosed)
7. Uncontrolled secondary hyperparathyroidism：PTH or iPTH>9×ULN；
8. History of malignancy within 5 years
9. Acute coronary syndrome, strokes (except for lacunar cerebral infarction), serious thromboembolism (eg. DVT or PE) within 6 months before the screening period
10. NYHA grade III or IV of congestive heart failure or severe arrythmia(including ventricular tachycardia, ventricular fibrillation, AV-block III etc.) within 6 months before screening
11. Pregnant or during lactation period or not willing to get contraception
12. Planning to receive renal transplantation within 2 months
13. Accepted blood transfusion within 3 months.
14. Serum ferritin，SF>500 μg/L
15. Planning to recieve the treatment as operations, chemotherapies or radiotherapies etc. during the research period
16. Other situations not suitable for inclusion decided by researchers. Rescreening is allowed if it failed in the first time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2027-02-09 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in hemoglobin concentration from baseline to week 8 | Screening period，Day 1，Week 1，Week 4，Week 8
  Full blood count

SECONDARY OUTCOMES:
Changes in hemoglobin concentration from baseline to week 4 | Screening period，Day 1，Week 1，Week 4
  Full blood count
Iron metabolism indices and reticulocyte count at week 8 | Screening period，Day 1，Week 1，Week 4，Week 8
  Iron metabolism indices and reticulocyte count
Iron metabolism indices and reticulocyte count at week 4 | Screening period，Day 1，Week 1，Week 4
  Iron metabolism indices and reticulocyte count
Compound cardiovascular adverse events at Week 8 | Through study completion, an average of 1 year
  Recording and observation with the reference of clinical symptoms and the results of EKG, NT-proBNP, cardiac troponin, CK-MB and myoglobin etc.
Adverse Events | Through study completion, an average of 1 year
  Recording and observation with the reference of clinical symptoms and the results of laboratory indices and other indices for safety

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalra PA, Bhandari S, Saxena S, Agarwal D, Wirtz G, Kletzmayr J, Thomsen LL, Coyne DW. A randomized trial of iron isomaltoside 1000 versus oral iron in non-dialysis-dependent chronic kidney disease patients with anaemia. Nephrol Dial Transplant. 2016 Apr;31(4):646-55. doi: 10.1093/ndt/gfv293. Epub 2015 Aug 6. PMID 26250435
- [Background] Bhandari S, Kalra PA, Kothari J, Ambuhl PM, Christensen JH, Essaian AM, Thomsen LL, Macdougall IC, Coyne DW. A randomized, open-label trial of iron isomaltoside 1000 (Monofer(R)) compared with iron sucrose (Venofer(R)) as maintenance therapy in haemodialysis patients. Nephrol Dial Transplant. 2015 Sep;30(9):1577-89. doi: 10.1093/ndt/gfv096. Epub 2015 Apr 28. PMID 25925701
- [Background] Bhandari S, Kalra PA, Berkowitz M, Belo D, Thomsen LL, Wolf M. Safety and efficacy of iron isomaltoside 1000/ferric derisomaltose versus iron sucrose in patients with chronic kidney disease: the FERWON-NEPHRO randomized, open-label, comparative trial. Nephrol Dial Transplant. 2021 Jan 1;36(1):111-120. doi: 10.1093/ndt/gfaa011. PMID 32049331
- [Background] Futterer S, Andrusenko I, Kolb U, Hofmeister W, Langguth P. Structural characterization of iron oxide/hydroxide nanoparticles in nine different parenteral drugs for the treatment of iron deficiency anaemia by electron diffraction (ED) and X-ray powder diffraction (XRPD). J Pharm Biomed Anal. 2013 Dec;86:151-60. doi: 10.1016/j.jpba.2013.08.005. Epub 2013 Aug 14. PMID 23998966
- [Background] Jahn MR, Andreasen HB, Futterer S, Nawroth T, Schunemann V, Kolb U, Hofmeister W, Munoz M, Bock K, Meldal M, Langguth P. A comparative study of the physicochemical properties of iron isomaltoside 1000 (Monofer), a new intravenous iron preparation and its clinical implications. Eur J Pharm Biopharm. 2011 Aug;78(3):480-91. doi: 10.1016/j.ejpb.2011.03.016. Epub 2011 Mar 23. PMID 21439379
- [Background] Auerbach M, Henry D, DeLoughery TG. Intravenous ferric derisomaltose for the treatment of iron deficiency anemia. Am J Hematol. 2021 Jun 1;96(6):727-734. doi: 10.1002/ajh.26124. Epub 2021 Feb 26. PMID 33580972
- [Background] Auerbach M, Gafter-Gvili A, Macdougall IC. Intravenous iron: a framework for changing the management of iron deficiency. Lancet Haematol. 2020 Apr;7(4):e342-e350. doi: 10.1016/S2352-3026(19)30264-9. PMID 32220343
- [Background] Bazeley JW, Wish JB. Recent and Emerging Therapies for Iron Deficiency in Anemia of CKD: A Review. Am J Kidney Dis. 2022 Jun;79(6):868-876. doi: 10.1053/j.ajkd.2021.09.017. Epub 2021 Nov 7. PMID 34758368
- [Background] Cancelo-Hidalgo MJ, Castelo-Branco C, Palacios S, Haya-Palazuelos J, Ciria-Recasens M, Manasanch J, Perez-Edo L. Tolerability of different oral iron supplements: a systematic review. Curr Med Res Opin. 2013 Apr;29(4):291-303. doi: 10.1185/03007995.2012.761599. Epub 2013 Feb 6. PMID 23252877
- [Background] Drueke TB, Parfrey PS. Summary of the KDIGO guideline on anemia and comment: reading between the (guide)line(s). Kidney Int. 2012 Nov;82(9):952-60. doi: 10.1038/ki.2012.270. Epub 2012 Aug 1. PMID 22854645
- [Background] Batchelor EK, Kapitsinou P, Pergola PE, Kovesdy CP, Jalal DI. Iron Deficiency in Chronic Kidney Disease: Updates on Pathophysiology, Diagnosis, and Treatment. J Am Soc Nephrol. 2020 Mar;31(3):456-468. doi: 10.1681/ASN.2019020213. Epub 2020 Feb 10. PMID 32041774
- [Background] Molnar MZ, Mehrotra R, Duong U, Kovesdy CP, Kalantar-Zadeh K. Association of hemoglobin and survival in peritoneal dialysis patients. Clin J Am Soc Nephrol. 2011 Aug;6(8):1973-81. doi: 10.2215/CJN.01050211. Epub 2011 Jul 22. PMID 21784829
- [Background] Li S, Foley RN, Collins AJ. Anemia, hospitalization, and mortality in patients receiving peritoneal dialysis in the United States. Kidney Int. 2004 May;65(5):1864-9. doi: 10.1111/j.1523-1755.2004.00584.x. PMID 15086928
- [Background] Horl WH. Anaemia management and mortality risk in chronic kidney disease. Nat Rev Nephrol. 2013 May;9(5):291-301. doi: 10.1038/nrneph.2013.21. Epub 2013 Feb 26. PMID 23438972
- [Background] Fishbane S, Spinowitz B. Update on Anemia in ESRD and Earlier Stages of CKD: Core Curriculum 2018. Am J Kidney Dis. 2018 Mar;71(3):423-435. doi: 10.1053/j.ajkd.2017.09.026. Epub 2018 Jan 11. PMID 29336855
- [Background] Cheng CK, Chan J, Cembrowski GS, van Assendelft OW. Complete blood count reference interval diagrams derived from NHANES III: stratification by age, sex, and race. Lab Hematol. 2004;10(1):42-53. PMID 15070217
- [Background] Yang C, Yang Z, Wang J, Wang HY, Su Z, Chen R, Sun X, Gao B, Wang F, Zhang L, Jiang B, Zhao MH. Estimation of Prevalence of Kidney Disease Treated With Dialysis in China: A Study of Insurance Claims Data. Am J Kidney Dis. 2021 Jun;77(6):889-897.e1. doi: 10.1053/j.ajkd.2020.11.021. Epub 2021 Jan 7. PMID 33421457
- [Background] GBD Chronic Kidney Disease Collaboration. Global, regional, and national burden of chronic kidney disease, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2020 Feb 29;395(10225):709-733. doi: 10.1016/S0140-6736(20)30045-3. Epub 2020 Feb 13. PMID 32061315